CLINICAL TRIAL: NCT03044717
Title: How Nutrition Education in Cardiology Fellows and Faculty Affects Clinical Practice Over a Six-Month Period
Brief Title: Nutrition Education in Fellows
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201700026
Record Dates: First submitted 2017-02-02; First posted 2017-02-07 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Medical Education
Keywords: Nutrition Education; Cardiology Fellows
MeSH Terms: interventions — Nutrition Surveys

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiology fellows and faculty: Fill out a nutrition survey three times at 0, 3, and 6 months and be present at a prevention educational conference every 5 weeks until the end of the study.
  This group will also complete a 3-hour nutrition module prior to study completion.
  Interventions: Other: Nutrition survey; Other: Educational Conference; Other: 3-hour nutrition module

INTERVENTIONS:
Other: Nutrition survey — Survey will be done prior to the initiation of the education
Other: Educational Conference — A prevention educational conference will be available to attend once every 5 weeks.
Other: 3-hour nutrition module — Nutrition module will be provided by the Gaples Institute to participants as part of this study. This will be completed online via e-mail
  Other Names: Nutrition module

SUMMARY:
The purpose of this research study is to assess comfort of cardiology fellows and faculty with nutrition and its role in cardiovascular disease and to determine if increasing education in this arena will change clinical practice.

DETAILED DESCRIPTION:
The aim of this project is to educate the fellows and faculty about nutrition. This will be done with a 3-hour nutrition module provided by the Gaples Institute. The Gaples Institute is a non-profit organization advocating natural strategies balanced with conventional medicine. The module will be provided free of charge for this education. There will also be a prevention education conference once every five weeks.

The secondary aim is to affect change in clinical practice among fellows and faculty. With an intensive nutrition education spanned over six months, the goal is to see if investigators can affect change in clinical practice. The nutrition module online will be available to those who participate in the study. The study participants are required to complete the 3-hour nutrition module prior to the six month completion of this study.

ELIGIBILITY:
Inclusion Criteria:

* All general cardiology fellow, faculty, internal medicine, residents, fellows will be asked to be part of this study.
* Male or females, 25 years or older

Exclusion Criteria:

* None

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiology fellow, faculty, internal medicine, residents, fellows
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2018-01-27 (Actual)

PRIMARY OUTCOMES:
Changes in behavior will be measured by method of Nutrition Survey | Change from Baseline, 3 months, and 6 months
  Nutrition Survey will be assessed at baseline, 3 months, and 6 months for changes in behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Aggarwal, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Survey data will be maintained on an electronic enrollment log created and maintained by research staff. The electronic enrollment log will be maintained on a secure institutional server and only accessible to research staff. When the project is closed, the enrollment log with identifiable information will be destroyed.